CLINICAL TRIAL: NCT07096713
Title: Evaluating the Efficacy and Safety of Brolucizumab Versus Aflibercept on Visual and Anatomical Outcomes in Diabetic Macular Edema: A Retrospective Comparative Study
Brief Title: Brolucizumab Versus Aflibercept on Visual and Anatomical Outcomes in Diabetic Macular Edema
Acronym: Anti-VEGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brolucizumab Vs Aflibercept
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2023-01

CONDITIONS: Anti-VEGF Therapy
Keywords: Diabetic macular edema; Brolucizumab; Aflibercept

STUDY DESIGN:
Intervention Model Description: This retrospective comparative cohort study aims to evaluate the efficacy and safety of intravitreal Brolucizumab versus Aflibercept in patients with center-involving diabetic macular edema (DME). A total of 38 eyes from 38 patients treated at Benha University Hospital between January 2023 and June 2024 were included. Patients were divided into two equal groups based on the anti-VEGF agent received: 19 eyes were treated with Brolucizumab 6 mg, and 19 eyes with Aflibercept 2 mg. The study compares visual acuity, central retinal thickness, number of injections, and adverse events over a 6-month follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Brolucizumab Group (Experimental): Description:
  This group included 19 eyes of 19 patients who received intravitreal Brolucizumab (6 mg/0.05 mL) injections for center-involving diabetic macular edema.
  Intervention Type: Drug
  Intervention Name: Brolucizumab 6 mg
  Dose/Frequency: Administered intravitreally as needed based on clinical evaluation
  Interventions: Drug: Intervention 1: Brolucizumab
- Arm 2: Aflibercept Group (Active Comparator): This group included 19 eyes of 19 patients who received intravitreal Aflibercept (2 mg/0.05 mL) injections for center-involving diabetic macular edema.
  Intervention Type: Drug
  Intervention Name: Aflibercept 2 mg
  Dose/Frequency: Administered intravitreally as needed based on clinical evaluation
  Interventions: Drug: Intervention 2: Aflibercept

INTERVENTIONS:
Drug: Intervention 1: Brolucizumab — Intravitreal injection of Brolucizumab (6 mg/0.05 mL) for the treatment of center-involving diabetic macular edema.
  Arms: Arm 1: Brolucizumab Group
Drug: Intervention 2: Aflibercept — Intravitreal injection of Aflibercept (2 mg/0.05 mL) for the treatment of center-involving diabetic macular edema.
  Arms: Arm 2: Aflibercept Group

SUMMARY:
This retrospective, comparative cohort study included 38 eyes from 38 patients with center-involving diabetic macular edema (DME), treated at Benha University Hospital. Patients were divided into two groups: 19 eyes received intravitreal Brolucizumab (6 mg), and 19 eyes received intravitreal Aflibercept (2 mg), with the aim of comparing their efficacy and safety over a 6-month period.

DETAILED DESCRIPTION:
The study retrospectively evaluated real-world outcomes of anti-VEGF therapy in treatment-naïve patients with center-involving DME. Participants were assigned into two equal groups based on the anti-VEGF agent received: Group A was treated with intravitreal Brolucizumab (6 mg), and Group B with intravitreal Aflibercept (2 mg). All patients underwent comprehensive ophthalmic evaluation at baseline and at monthly intervals, including best-corrected visual acuity (BCVA) assessment and optical coherence tomography (OCT) to monitor central retinal thickness (CRT). The primary outcomes were changes in BCVA and CRT from baseline to 6 months, while secondary outcomes included the number of injections received and any adverse events. This study aimed to provide comparative insights into the efficacy, anatomical response, and safety profile of the two anti-VEGF agents in managing DME in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with center-involving diabetic macular edema (DME) confirmed by spectral-domain optical coherence tomography (SD-OCT).
* Central macular thickness (CMT) > 350 µm at baseline.
* Treatment-naïve patients (no prior intravitreal injections or laser therapy for DME).

Exclusion Criteria:

* Patients with media opacity (e.g., corneal opacities, dense vitreous hemorrhage).
* Significant cataract affecting visual acuity or OCT imaging quality.
* Traction maculopathy or vitreomacular traction.
* Central macular thickness < 350 µm at baseline.
* History of vasculitis or autoimmune diseases (e.g., systemic lupus erythematosus [SLE]).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) from Baseline to 6 Months | Baseline and 6 months
  Measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart or Snellen equivalent, converted to logMAR. The primary measure is the mean change in BCVA after treatment with either Brolucizumab or Aflibercept.
Change in Central Retinal Thickness (CRT) from Baseline to 6 Months | Baseline and 6 months
  Assessed by spectral-domain optical coherence tomography (SD-OCT). The outcome is the mean change in CRT in micrometers, reflecting anatomical response to treatment.

SECONDARY OUTCOMES:
Total Number of Intravitreal Injections Over 6 Months | From baseline to month 6
  The cumulative number of injections each patient received, to compare treatment burden between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banha, Cairo Governorate, Egypt